

#### **MIDAS Quality Enhancement Research Initiative**

Center for Clinical Management Research 2215 Fuller Rd (152) Ann Arbor, MI 48109 (734) 845-3502

Official Title of Project: Maintaining Implementation Through Dynamic Adaptations (MIDAS) - Suicide

Prevention 2.0 Clinical Telehealth (SP 2.0)

ClinicalTrials.gov ID: NCT06011759

Date: 10/24/2025

## **Background**

The suicide rate for Veterans is significantly greater than among non-Veteran U.S. adults. According to the VA Office of Suicide Prevention's 2024 National Veteran Suicide Prevention Annual Report, there were 6,407 Veteran suicide deaths in 2022 and suicide is the second leading cause of death for Veterans under 45 years old. To improve access to effective suicide prevention treatments, the Veterans Health Administration (VHA) recently initiated the Suicide Prevention 2.0 Clinical Telehealth (SP 2.0) program; a regional hub model for virtually delivering evidence-based suicide-specific psychotherapies. Referrals to SP 2.0 vary widely across VHA facilities. This study's aim was to identify barriers and facilitators for program referrals to inform program and facility leaders and the deployment of implementation strategies.

SP 2.0 Clinical Telehealth operates Clinical Resource Hubs at the VISN level and uses evidence-based interventions for suicide prevention, such as Safety Planning Intervention, Cognitive Behavioral Therapy for Suicide Prevention, Problem Solving Therapy for Suicide Prevention, and Dialectical Behavior Therapy.

1. Morral et al., 2023, <a href="https://doi.org/10.1001/jamanetworkopen.2023.24191">https://doi.org/10.1001/jamanetworkopen.2023.24191</a>

This project will include test two implementation strategies: (1) academic detailing (AD) and (2) Learn. Engage. Act. Process. (LEAP) team-based quality improvement (QI). The first strategy, AD, is designed to provide individual providers with the knowledge and motivation to use the EBPs. The second implementation strategy, LEAP, is a team-based strategy that engages frontline providers and staff in incremental cycles of improvement in the use of the EBP with the support of a coach. The LEAP program provides coaching within a structured, paced curriculum over a 6-month period, during which teams complete one improvement project following a Plan-Do-Study-Act (PDSA) cycle of change.<sup>2</sup>

2. Damschroder et al., 2022, https://doi.org/10.1186/s43058-022-00297-z

### **Aims**

This study will evaluate the following aims:

- 1. Compare the effectiveness of two implementation strategies, LEAP Quality Improvement Learning Program and Academic Detailing (AD), on the following outcomes:
  - a. SP2Clin Metric (primary outcome) The quarterly SP2Clin metric data is reported and available on a VA national dashboard. The SP2Clin metric is calculated by the number of suicide prevention telehealth consults submitted among those with a suicide behavior event.

- b. Referral to SP 2.0 Clinic (secondary outcome) Change in number of referrals to the Suicide Prevention 2.0 Clinical Telehealth (SP 2.0) initiative
- 2. We will also examine other pre-specified outcomes related to the implementation strategies:
  - a. Change in quality improvement skills application a 16-item measure of change in quality improvement skills application. Values 1 to 4 where higher values indicate more frequent use of quality improvement skills.
  - b. Provider satisfaction with academic detailing 7 items measuring satisfaction with Academic Detailing. Each response option uses a Likert-type scale with values 1 to 5 where higher values indicate higher satisfaction.
  - c. Provider satisfaction with LEAP 6-item measure of satisfaction with LEAP. Values 1 to 5 where higher values indicate higher satisfaction

#### Methods

Interested sites will be provided a site orientation meeting that outlines details around study participation and the QI strategies being offered. In prior trials, we found that random assignment into QI strategies (LEAP and/or AD) was a barrier to participation due to time constraints and limited staff bandwidth. For this study, we will allow sites to elect which QI strategies they would like to participate in based on their individual site characteristics, including site-specific barriers and facilitators. We will also engage both front-line workers and leadership during site recruitment to ensure leadership supports front-line workers' participation in the project.

# **Outcomes and Analysis**

To examine the effect of engagement in quality improvement activity on referral to the SP 2.0 program, we will compare participating sites with similar non-participating sites. Non-participating sites will be selected as matched controls, one for each participating site. Control sites will be matched 1:1 to participating sites on number of suicide behavior events and prevalence of Suicide Prevention Telehealth Program consults submitted at baseline. T-tests will be conducted to compare participating and control sites on the primary and secondary outcomes. For the other pre-specified outcomes, descriptive statistics will be generated.

#### **List of Abbreviations**

Academic detailing (AD)

Learn. Engage. Act. Process. (LEAP)

Maintaining Implementation through Dynamic Adaptations (MIDAS)

Plan-Do-Study-Act (PDSA)

Quality improvement (QI)

Suicide Prevention 2.0 Clinical Telehealth (SP 2.0)